CLINICAL TRIAL: NCT00624052
Title: An Open Label Trial of the Efficacy and Safety of Chronic Administration of the Fixed Dose Combination of Telmisartan 40mg + Amlodipine 10mg or Fixed Dose Combination of Telmisartan 80mg + Amlodipine 10mg Tablets Alone or in Combination With Other Antihypertensive Medications in Patients With Hypertension
Brief Title: 26-week Open Study of telmisartan40mg+amlodipine10mg or telmisartan80mg+amlodipine10 mg in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 1235.8
Record Dates: First submitted 2008-02-05; First posted 2008-02-26 (Estimated); Results first posted 2010-03-25 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

INTERVENTIONS:
Drug: fixed-dose combination of telmisartan 40mg+amlodipine 10mg
Drug: fixed-dose combination of telmisartan 80mg+amlodipine10mg

SUMMARY:
The primary objective of this trial is to assess the efficacy and safety of the fixed dose combinations telmisartan 40mg/amlodipine 10mg (T40/A10) or telmisartan 80mg/amlodipine 10mg (T80/A10) during open-label treatment for at least six months.

An additional objective is to assess the efficacy and safety of concomitant administration of either T40/A10 or T80/A10 with any other therapies commonly used in the treatment of hypertension.

The primary endpoint is the proportion of patients achieving DBP control (defined as mean seated DBP < 90 mmHg at trough i.e. approximately 24 hours after last dose of study treatment) at six months of treatment or at last trough observation during the treatment period (i.e. last trough observation carried forward).

ELIGIBILITY:
Inclusion Criteria:

- diagnosis of essential hypertension

Exclusion Criteria:

* pregnancy, breast-feeding, unwilling to use effective contraception (if female of child-bearing potential).
* development of any condition in the preceding trial that could be worsened by telmisartan 40mg/amlodipine 10mg (T40/A10) or telmisartan 80mg/amlodipine 10mg (T80/A10).
* discontinuation from the preceding trial.
* known or suspected secondary hypertension.
* mean seated systolic blood pressure (SBP) >= 180 mmHg and/or mean seated diastolic blood pressure (DBP) >= 120 mmHg at any visit.
* any clinically significant hepatic impairment or severe renal impairment bilateral renal artery stenosis or renal artery stenosis in a solitary kidney or post post-renal transplant.
* clinically relevant hyperkalaemia.
* uncorrected volume or sodium depletion.
* primary aldosteronism.
* hereditary fructose or lactose intolerance.
* symptomatic congestive heart failure.
* patients who have previously experienced symptoms characteristic of angioedema during treatment with angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs).
* any new drug or alcohol dependency since signing consent of the preceding trial.
* concurrent participation in another clinical trial or any investigational therapy since completing the preceding trial.
* hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve.
* known allergic hypersensitivity to any component of the formulations under investigation. [Includes known hypersensitivity to telmisartan or other ARBs or amlodipine or other dihydropyridine calcium channel blockers (CCBs).] non-compliance with study medication (defined as <80% or >120%) during the preceding trial.
* administration of ARBs or dihydropyridine CCBs (apart from trial medication). any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of telmisartan and amlodipine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 838 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (92):
- Australia (5):
  - 1235.8.61003 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 1235.8.61004 Boehringer Ingelheim Investigational Site, Liverpool, New South Wales
  - 1235.8.61002 Boehringer Ingelheim Investigational Site, Kippa-Ring, Queensland
  - 1235.8.61001 Boehringer Ingelheim Investigational Site, Milton, Queensland
  - 1235.8.61005 Boehringer Ingelheim Investigational Site, Elizabeth Vale, South Australia
- Austria (5):
  - 1235.8.43007 Boehringer Ingelheim Investigational Site, Eggenburg
  - 1235.8.43006 Boehringer Ingelheim Investigational Site, Hainburg A.d. Donau
  - 1235.8.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1235.8.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 1235.8.43003 Boehringer Ingelheim Investigational Site, Vienna
- Bulgaria (9):
  - 1235.8.35912 Boehringer Ingelheim Investigational Site, Burgas
  - 1235.8.35902 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.8.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.8.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.8.35905 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.8.35906 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.8.35907 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.8.35910 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.8.35911 Boehringer Ingelheim Investigational Site, Sofia
- Czechia (7):
  - 1235.8.42002 Boehringer Ingelheim Investigational Site, Benátky nad Jizerou
  - 1235.8.42006 Boehringer Ingelheim Investigational Site, Brno
  - 1235.8.42001 Boehringer Ingelheim Investigational Site, Pilsen
  - 1235.8.42003 Boehringer Ingelheim Investigational Site, Prague
  - 1235.8.42004 Boehringer Ingelheim Investigational Site, Příbram
  - 1235.8.42005 Boehringer Ingelheim Investigational Site, Slaný
  - 1235.8.42007 Boehringer Ingelheim Investigational Site, Strakonice
- Ireland (5):
  - 1235.8.35304 Boehringer Ingelheim Investigational Site, Birr
  - 1235.8.35305 Boehringer Ingelheim Investigational Site, Carrigtowhill
  - 1235.8.35303 Boehringer Ingelheim Investigational Site, Gorey, Co. Wexford
  - 1235.8.35306 Boehringer Ingelheim Investigational Site, Mallow
  - 1235.8.35301 Boehringer Ingelheim Investigational Site, New Ross
- Italy (3):
  - 1235.8.39002 Boehringer Ingelheim Investigational Site, Broni (pv)
  - 1235.8.39006 Boehringer Ingelheim Investigational Site, Coppito (AQ)
  - 1235.8.39001 Boehringer Ingelheim Investigational Site, Ferrara
- New Zealand (3):
  - 1235.8.64003 Boehringer Ingelheim Investigational Site, Dunedin
  - 1235.8.64002 Boehringer Ingelheim Investigational Site, Otahuhu, Auckland
  - 1235.8.64001 Boehringer Ingelheim Investigational Site, Tauranga
- Russia (9):
  - 1235.8.70004 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.8.70005 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.8.70006 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.8.70007 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.8.70008 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.8.70009 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.8.70010 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.8.70011 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.8.70012 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (7):
  - 1235.8.42103 Boehringer Ingelheim Investigational Site, Dolný Kubín
  - 1235.8.42106 Boehringer Ingelheim Investigational Site, Kralovsky Chmlec
  - 1235.8.42104 Boehringer Ingelheim Investigational Site, Liptovský Mikuláš
  - 1235.8.42102 Boehringer Ingelheim Investigational Site, Považská Bystrica
  - 1235.8.42105 Boehringer Ingelheim Investigational Site, Prešov
  - 1235.8.42101 Boehringer Ingelheim Investigational Site, Trenčín
  - 1235.8.42107 Boehringer Ingelheim Investigational Site, Vráble
- Spain (11):
  - 1235.8.34008 Boehringer Ingelheim Investigational Site, Badalona
  - 1235.8.34010 Boehringer Ingelheim Investigational Site, Badalona
  - 1235.8.34009 Boehringer Ingelheim Investigational Site, Barcelona
  - 1235.8.34001 Boehringer Ingelheim Investigational Site, Jerez de La Frontera (Cádiz)
  - 1235.8.34006 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1235.8.34003 Boehringer Ingelheim Investigational Site, Madrid
  - 1235.8.34004 Boehringer Ingelheim Investigational Site, Madrid
  - 1235.8.34012 Boehringer Ingelheim Investigational Site, Mataró
  - 1235.8.34002 Boehringer Ingelheim Investigational Site, Oviedo
  - 1235.8.34005 Boehringer Ingelheim Investigational Site, Santa Coloma de Gramanet
  - 1235.8.34011 Boehringer Ingelheim Investigational Site, Santa Coloma de Gramanet
- Ukraine (13):
  - 1235.8.38010 Boehringer Ingelheim Investigational Site, Dnipro
  - 1235.8.38001 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.8.38003 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.8.38008 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.8.38011 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.8.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.8.38006 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.8.38012 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.8.38013 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.8.38002 Boehringer Ingelheim Investigational Site, Lviv
  - 1235.8.38005 Boehringer Ingelheim Investigational Site, Odesa
  - 1235.8.38009 Boehringer Ingelheim Investigational Site, Odesa
  - 1235.8.38007 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (15):
  - 1235.8.44010 Boehringer Ingelheim Investigational Site, Bexhill-on-Sea
  - 1235.8.44008 Boehringer Ingelheim Investigational Site, Blackpool
  - 1235.8.44016 Boehringer Ingelheim Investigational Site, Blackpool
  - 1235.8.44011 Boehringer Ingelheim Investigational Site, Burbage
  - 1235.8.44007 Boehringer Ingelheim Investigational Site, Chestfield, Whitstable
  - 1235.8.44005 Boehringer Ingelheim Investigational Site, Chorley
  - 1235.8.44002 Boehringer Ingelheim Investigational Site, Edgbaston, Birmingham
  - 1235.8.44009 Boehringer Ingelheim Investigational Site, Ely
  - 1235.8.44001 Boehringer Ingelheim Investigational Site, Fowey
  - 1235.8.44003 Boehringer Ingelheim Investigational Site, Glasgow
  - 1235.8.44012 Boehringer Ingelheim Investigational Site, Penzance
  - 1235.8.44013 Boehringer Ingelheim Investigational Site, Plymouth
  - 1235.8.44004 Boehringer Ingelheim Investigational Site, Reading
  - 1235.8.44015 Boehringer Ingelheim Investigational Site, St Austell
  - 1235.8.44006 Boehringer Ingelheim Investigational Site, Whitstable

REFERENCES:
- [Derived] Neldam S, Edwards C, Lang M, Jones R; TEAMSTA-5 and TEAMSTA-10 Investigators. Long-Term Tolerability and Efficacy of Single-Pill Combinations of Telmisartan 40-80 mg Plus Amlodipine 5 or 10 mg in Patients Whose Blood Pressure Was Not Initially Controlled by Amlodipine 5-10 mg: Open-Label, Long-Term Follow-Ups of the TEAMSTA-5 and TEAMSTA-10 Studies. Curr Ther Res Clin Exp. 2012 Feb;73(1-2):65-84. doi: 10.1016/j.curtheres.2012.02.004. PMID 24653513

RESULTS

PARTICIPANT FLOW:
Groups:
- Telmisartan 40mg and Amlodipine 10mg: Patients who were randomised to telmisartan 40mg and amlodipine 10mg and were on this dose at their last study visit
- Randomised Telmisartan 80mg and Amlodipine 10mg: Patients who were randomised to telmisartan 80mg and amlodipine 10mg and were on this dose at their last study visit
- Titrated Telmisartan 80mg and Amlodipine 10mg: Patients who were randomised to telmisartan 40mg and amlodipine 10mg but were titrated to telmisartan 80mg and amlodipine 10mg and were on this dose at their last study visit
- Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on: Patients who were on either telmisartan 40 mg or 80mg and amlodipine 10mg plus another antihypertensive medication at their last study visit
Period: Overall Study
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Started | 219 | 436 | 91 | 92
Completed | 204 | 422 | 88 | 88
Not Completed | 15 | 14 | 3 | 4
Not completed — Adverse Event | 7 | 6 | 0 | 3
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 1 | 0
Not completed — Non compliant with the protocol | 2 | 1 | 1 | 1
Not completed — Consent withdrawn | 3 | 1 | 1 | 0
Not completed — Changed job/ran out if meds | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on | Total
Number analyzed (Participants) | 219 | 436 | 91 | 92 | 838
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (9.9) | 57.3 (9.4) | 55.2 (9.7) | 53.3 (10.3) | 56.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 206 | 31 | 37 | 367
  Male | 126 | 230 | 60 | 55 | 471

OUTCOME MEASURES:

1. Primary Outcome: Trough Seated Diastolic Blood Pressure (DBP) Control
Description: The number of patients who reached the target DBP of <90mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: The full analysis set of patients. All patients who took at least one dose of study medication and have at least one on treatment BP measurement 20-30 hours post dose
Measure: Number; unit: patients
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 216 | 436 | 91 | 92
patients
  Yes (DBP<90 mmHg) | 201 | 402 | 72 | 70
  No (DBP>=90 mmHg) | 15 | 34 | 19 | 22
Statistical Analysis 1: Comparison: Telmisartan 40mg and Amlodipine 10mg vs Randomised Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI [0.47 to 1.66]
Statistical Analysis 2: Comparison: Telmisartan 40mg and Amlodipine 10mg vs Titrated Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.28, 95% CI [0.14 to 0.59]
Statistical Analysis 3: Comparison: Telmisartan 40mg and Amlodipine 10mg vs Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.24, 95% CI [0.12 to 0.48]
Statistical Analysis 4: Comparison: Randomised Telmisartan 80mg and Amlodipine 10mg vs Titrated Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.32, 95% CI [0.17 to 0.59]
Statistical Analysis 5: Comparison: Randomised Telmisartan 80mg and Amlodipine 10mg vs Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.27, 95% CI [0.15 to 0.49]
Statistical Analysis 6: Comparison: Titrated Telmisartan 80mg and Amlodipine 10mg vs Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI [0.42 to 1.68]

2. Secondary Outcome: Trough Seated Systolic Blood Pressure (SBP) Control
Description: The number of patients who reached the target SBP of >=140mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 216 | 436 | 91 | 92
patients
  Yes (SBP<140 mmHg) | 179 | 366 | 70 | 51
  No (SBP>=140 mmHg) | 37 | 70 | 21 | 41

3. Secondary Outcome: Change From Baseline to End of Study in Trough Seated Diastolic Blood Pressure
Description: Change from baseline to the end of study in trough DBP. Baseline is defined as visit 3 of trial 1235.6
Time Frame: Baseline is defined as visit 3 of study NCT00553267 and end of study as 34 weeks or last value on treatment
Population: All patients who took at least one dose of study medication, have a trough baseline measurement (Visit 3 NCT00553267) and at least one on treatment BP measurement 20-30 hours post dose
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 214 | 434 | 87 | 91
mmHg | -13.41 (0.44) | -13.36 (0.31) | -11.52 (0.69) | -10.64 (0.67)

4. Secondary Outcome: Change in DBP From Last Available Trough in NCT00553267 to Last Available Trough in NCT00624052
Description: The difference between the last available troughs represents the additional reduction in DBP in this study
Time Frame: Last available trough in NCT00553267 to end of study (34 weeks or last value on treatment)
Population: All patients who took at least one dose of study medication, have a trough end of study measurement from NCT00553267 and at least one on treatment BP measurement 20-30 hours post dose
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 213 | 430 | 91 | 92
mmHg | -4.36 (0.48) | -4.97 (0.34) | -5.51 (0.74) | -5.43 (0.73)

5. Secondary Outcome: Change From Baseline to End of Study in Trough Seated Systolic Blood Pressure
Description: Change from baseline to the end of study in trough SBP. Baseline is defined as visit 3 of trial 1235.6
Time Frame: Baseline is defined as visit 3 of study NCT00553267 and end of study as 34 weeks or last value on treatment
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 214 | 434 | 87 | 91
mmHg | -14.76 (0.72) | -15.93 (0.5) | -14.85 (1.12) | -12.44 (1.1)

6. Secondary Outcome: Change in SBP From Last Available Trough in NCT00553267 to Last Available Trough in NCT00624052
Description: The difference between the last available troughs represents the additional reduction in SBP in this study
Time Frame: Last available trough in NCT00624052 to end of study (34 weeks or last value on treatment)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 213 | 430 | 91 | 92
mmHg | -4.73 (0.73) | -6.02 (0.51) | -6.55 (1.11) | -5.61 (1.1)

7. Secondary Outcome: Trough Seated DBP Response
Description: The number of patients who reach the target DBP of <90mmHg or had a reduction in DBP >= 10mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: All patients who took at least one dose of study medication, have a trough baseline measurement (Visit 3 NCT 00553267) and at least one on treatment BP measurement 20-30 hours post dose
Measure: Number; unit: patients
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 214 | 434 | 87 | 91
patients
  Yes (Responder) | 201 | 405 | 71 | 73
  No (Non-responder) | 13 | 29 | 16 | 18

8. Secondary Outcome: Trough Seated SBP Response
Description: The number of patients who reach the target SBP of <140mmHg or had a reduction in SBP >= 15 mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: as for outcome 7
Measure: Number; unit: patients
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 214 | 434 | 87 | 91
patients
  Yes (Responder) | 190 | 401 | 75 | 69
  No (Non-responder) | 24 | 33 | 12 | 22

9. Secondary Outcome: Trough BP Normality Classes
Description: The number of patients who reach predefined BP categories
Time Frame: End of study (34 weeks or last value on treatment)
Measure: Number; unit: patients
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Randomised Telmisartan 80mg and Amlodipine 10mg | Titrated Telmisartan 80mg and Amlodipine 10mg | Telmisartan 40mg or 80mg and Amlodipine 10mg + add-on
Number analyzed (Participants) | 213 | 430 | 91 | 92
patients
  Optimal (SBP<120 and DBP<80 mmHg) | 12 | 20 | 5 | 3
  Normal (SBP<130 and DBP<85 mmHg and not optimal) | 70 | 146 | 14 | 13
  High-normal (SBP<140 DBP<90 mmHg and not normal) | 94 | 189 | 46 | 29
  Stage 1 hypertension (SBP<160 and DBP<100 mmHg | 32 | 76 | 23 | 43
  Stage 2 hypertension (SBP>=160 and DBP>=100 mmHg) | 8 | 5 | 3 | 4

10. Secondary Outcome: Time to First Additional Antihypertensive
Description: Time from first intake of medication to first intake of an antihypertensive other than the study drug
Time Frame: up to 34 weeks
Population: The total of the number of patients in the BP normality classes. Decision to treat with additional antihypertensive was at investigator discretion. Some patients may have been deemed to be at higher cardiovascular risk therefore requiring additional antihypertensive treatment
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Telmisartan 40mg and Amlodipine 10mg
Number analyzed (Participants) | 121
Days | 91.9 (45.2)

11. Secondary Outcome: Number of Patients Requiring Additional Antihypertensive Therapy to Achieve DBP Control
Description: The number of patients with DBP control (DBP>=90 mmHg). Last trough DBP measurement before taking additional antihypertensive compared to last trough DBP taken on treatment
Time Frame: up to 34 weeks
Population: Decision to treat with additional antihypertensive was at investigator discretion. Some patients may have been deemed to be at higher cardiovascular risk therefore requiring additional antihypertensive treatment
Measure: Number; unit: patients
Arm/Group | Pre-antihypertensive: Yes (DBP<90 mmHg) | Pre-antihypertensive: No (DBP>=90 mmHg) | Pre-antihypertensive: Total
Number analyzed (Participants) | 31 | 90 | 121
patients
  Post-antihypertensive: Yes (DBP<90 mmHg) | 27 | 67 | 94
  Post-antihypertensive: No (DBP>=90 mmHg) | 4 | 23 | 27
  Post-antihypertensive: Total | 31 | 90 | 121

12. Secondary Outcome: Additional Reduction in DBP by Use of Additional Antihypertensive Therapy
Description: Difference in trough DBP from last visit before add-on therapy and last visit during NCT00624052
Time Frame: up to 34 weeks
Population: Total for the full analysis set. Decision to treat with additional antihypertensive was at investigator discretion. Some patients may have been deemed to be at higher cardiovascular risk therefore requiring additional antihypertensive treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 10mg
Number analyzed (Participants) | 121
mmHg | -6.79 (7.39)

13. Secondary Outcome: Additional Reduction in SBP by Use of Additional Antihypertensive Therapy
Description: Difference in trough SBP from last visit before add-on therapy and last visit during NCT00624052
Time Frame: up to 34 weeks
Population: Total for the full analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 10mg
Number analyzed (Participants) | 121
mmHg | -7.79 (12.37)

14. Secondary Outcome: Trough DBP Control Pre- and Post- Uptitration
Description: The number of patients with DBP control (DBP<90 mmHg). Last trough DBP measurement before uptitration to telmisartan 80mg and amlodipine 10mg compared to first trough DBP taken after uptitration. Uptitration could be based DBP>90 or investigator opinion.
Time Frame: up to 34 weeks
Population: 91 is the number of patients titrated to telmisartan 80mg. To get 582 you need to consider the randomised to telmisartan 80 mg patients and those with additional antihypertensive that were on telmisartan 80mg.
Measure: Number; unit: patients
Arm/Group | Pre-titration: Yes (DBP<90 mmHg) | Pre-titration: No (DBP>=90 mmHg) | Pre-titration: Total
Number analyzed (Participants) | 324 | 258 | 582
patients
  Post-titration: Yes (DBP<90 mmHg) | 306 | 168 | 474
  Post-titration: No (DBP>=90 mmHg) | 18 | 90 | 108
  Post-titration: Total | 324 | 258 | 582

ADVERSE EVENTS:
Time Frame: From day of first dose through to the day after last dose
Description: Safety data was analysed based upon actual dose of telmisartan and amlodipine the patient was on at the onset of AE regardless of additional antihypertensive
Groups:
- Telmisartan 40mg and Amlodipine 10mg: The 838 participants in the telmisartan 40mg/amlodipine 10mg group includes all participants
- Telmisartan 80mg and Amlodipine 10mg: The 611 participants in the telmisartan 80mg/amlodipine 10mg (T80/A10) group include 436 patients in the randomised T80/A10 group + 91 patients in the uptitrated T80/A10 group + XX patients in the T80/A10 + add-on group
Arm/Group | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Serious Adverse Events (participants affected / at risk) | 4/838 | 13/611
Other Adverse Events (participants affected / at risk) | 0/838 | 0/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40mg and Amlodipine 10mg (N=838) | Telmisartan 80mg and Amlodipine 10mg (N=611)
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Stent related infection (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Parasoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.